CLINICAL TRIAL: NCT00781495
Title: Determinants of Insulin-induced Weight Gain in Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Prof. dr. C. J. Tack, Radboud University Nijmegen Medical Centre
Other Study IDs: T2DM_insulin_weight gain
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes Mellitus; Weight Gain
Keywords: insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Gain; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- type 2 diabetes mellitus
  Interventions: Device: Sensewear Bodymedia armband

INTERVENTIONS:
Device: Sensewear Bodymedia armband — To assess physical activity levels patients will wear Sensewear bodymedia armband
  Other Names: Sensewear Bodymedia system

SUMMARY:
The purpose of this study is to find determinants of insulin-induced weight gain in type 2 diabetes mellitus

Primary objective: To find an association between weight gain after start of insulin therapy and physical activity levels.

DETAILED DESCRIPTION:
Insulin therapy is frequently needed to achieve adequate glycaemic control in type 2 diabetes mellitus (T2DM), but often at the expense of weight gain. Insulin-induced weight gain is obviously undesirable in an already overweight population and may negatively affect blood pressure, lipid levels, inflammatory and fibrinolytic parameters, adipocytokines and also deter further optimization of insulin therapy. It is unknown what determinants predict insulin-induced weight gain in type 2 diabetes mellitus.

The aim of this study therefore, is to assess determinants of insulin-induced weight gain in type 2 diabetes mellitus. In a retrospective and cross-sectional study (Jansen HJ et al., submitted) two extreme subgroups were identified (subjects with a weight gain above 80th percentile) and subgroup non-weight gainers (subjects with a weight gain below the 20th percentile). It was found that the gainers had less energy expenditure after initiation of insulin therapy than non-weight gainers. Therefore, the primary aim of this study is to detect an association between energy expenditure and weight gain

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes mellitus
* age 18-85 years
* Hba1c at baseline < 12.0%
* written informed consent

Exclusion Criteria:

* Clinical evidence of psychiatric, renal, cardiovascular or liver or other diseases which may influence study results regarding glucose and weight
* Patients with hormonal disorders which may influence weight (i.e. thyroid diseases), even if properly treated with stable hormonal levels
* Excessive alcohol consumption (>20 g/day), and drug abuse
* Use of thiazolidinedione derivatives (TZDs)
* Pregnancy or intention to become pregnant during the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus, selected from the out-patient clinic of the Radboud University Nijmegen Medical Centre and four other non-academic hospitals.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To detect an association between insulin-induced weight gain and physical activity levels | 1 year

SECONDARY OUTCOMES:
To assess the relationship between insulin-induced weight gain and cardiovascular risk profile | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Henry Jansen, MD, Principal Investigator — Radboud University Medical Center; Cees Tack, Prof.dr., Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant

REFERENCES:
- [Derived] Jansen HJ, Stienstra R, van Diepen JA, Hijmans A, van der Laak JA, Vervoort GM, Tack CJ. Start of insulin therapy in patients with type 2 diabetes mellitus promotes the influx of macrophages into subcutaneous adipose tissue. Diabetologia. 2013 Dec;56(12):2573-81. doi: 10.1007/s00125-013-3018-6. Epub 2013 Sep 25. PMID 24065152